CLINICAL TRIAL: NCT00298025
Title: A Phase IV, Multicenter, Open-label, Randomized Study to Compare the Safety and Efficacy of Cetrotide® 3 mg Versus Antagon™ in the Inhibition of a Premature LH Surge in a r-hFSH/hMG Stimulation Cycle With OCP Programming in Women Undergoing Ovarian Stimulation Prior to ART
Brief Title: A Study to Compare the Safety and Efficacy of Cetrotide® 3 Milligram (mg) Versus Antagon™ in Women Undergoing Ovarian Stimulation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: EMD Serono (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 24688
Record Dates: First submitted 2006-02-27; First posted 2006-03-01 (Estimated); Last update posted 2014-03-26 (Estimated); Status verified 2014-03

CONDITIONS: Infertile Women Undergoing Assisted Reproductive Technology (ART)
Keywords: Infertility; Cetrotide; Antagon; Recombinant human follicle stimulating hormone (r-hFSH); Human Menopausal Gonadotropin (hMG); Recombinant Human Choriogonadotropin (r-hCG)
MeSH Terms: conditions — Infertility | interventions — cetrorelix; ganirelix; Glycoprotein Hormones, alpha Subunit; follitropin alfa; Menotropins; Ovidrel; Chorionic Gonadotropin

ARMS (2):
- Cetrotide® (Experimental)
  Interventions: Drug: Cetrotide®; Drug: Recombinant human follicle stimulating hormone (r-hFSH); Drug: Human Menopausal Gonadotropin (hMG); Drug: Recombinant Human Choriogonadotropin (r-hCG)
- Antagon ™ (Active Comparator)
  Interventions: Drug: Antagon ™; Drug: Recombinant human follicle stimulating hormone (r-hFSH); Drug: Human Menopausal Gonadotropin (hMG); Drug: Recombinant Human Choriogonadotropin (r-hCG)

INTERVENTIONS:
Drug: Cetrotide® — Cetrotide® will be administered subcutaneously as 3 mg injection when the lead follicle is >=14 mm till r-hCG day. If the subject did not achieve follicular maturation and did not receive r-hCG within 4 days, then the Cetrotide® will be administered at dose of 0.25 mg subcutaneously on successive days until r-hCG day.
  Other Names: Cetrorelix acetate
  Arms: Cetrotide®
Drug: Antagon ™ — Antagon™ will be administered subcutaneously at a dose of 0.25 mg once daily when the lead follicle is >=14 mm until r-hCG day.
  Other Names: Ganirelix acetate
  Arms: Antagon ™
Drug: Recombinant human follicle stimulating hormone (r-hFSH) — Recombinant human follicle stimulating hormone (r-hFSH) will be administered at a starting dose of 225 international unit (IU) subcutaneously once daily from S1 up to Stimulation Day 5 (S5). Beginning on Stimulation Day 6 (S6), the r-hFSH dose will be individualized to the subject. The minimum and maximum daily doses are 75 IU and 450 IU, respectively until r-hCG day.
  Other Names: Gonal-f®
Drug: Human Menopausal Gonadotropin (hMG) — Human menopausal gonadotropin (hMG) will be administered subcutaneously daily at a dose of 75 IU till r-hCG day. The total daily dose of r-hFSH and hMG combined is not to exceed 450 IU (375 IU r-hFSH and 75 IU hMG).
  Other Names: Pergonal®
Drug: Recombinant Human Choriogonadotropin (r-hCG) — The r-hCG will be administered as a single dose of 250 microgram (mcg) subcutaneously when there is at least one follicle of >=18 mm and two additional follicles of >=16 mm with an appropriate plasma estradiol levels for the number and size of the existing follicles. The r-hCG will be administered within 36 hours after the last dose of the r-hFSH/hMG.
  Other Names: Ovidrel®; Choriogonadotropin alfa

SUMMARY:
To demonstrate the comparative safety and efficacy of Cetrotide® 3 milligram (mg) and Antagon™ in the inhibition of a premature luteinizing hormone (LH) surge in women undergoing ovarian stimulation with recombinant human follicle stimulating hormone/human menopausal gonadotropin (r-hFSH/hMG) prior to assisted reproductive technology (ART) and utilizing oral contraceptives pill (OCP) for cycle programming.

ELIGIBILITY:
Inclusion Criteria:

* Infertile women wishing to conceive whose physician had recommended that she can undergo ART
* Aged 18-39 years (inclusive)
* Regular menstrual cycles every 25-35 days
* Body mass index (BMI) less than 35 kilogram per square meter (kg/m^2)
* Has a transvaginal pelvic ultrasound scan within 6 weeks prior to OCP administration, as well as an Hysterosalpingography (HSG) or hysterosonogram or hysteroscopy within three years prior to OCP administration showing no clinically significant pelvic and/or uterine abnormality, which, in the Investigator's opinion, could impair ovarian response, embryo implantation or pregnancy continuation
* Normal cervical cytology, documented by Pap Smear, within six months prior to OCP administration
* If the subject had prior stimulation cycles, at least a 60-day washout period is required after the last dose of gonadotropin or clomiphene citrate; a 60-day washout is required after the last dose of Lupron® or Lupron Depot® 1-month; a 180-day washout period is required after the last dose of treatment with Depo-Provera® and Lupron Depot® 6-month; a 60-day washout is required after the last dose of oral contraceptives prior to OCP administration in the study
* Screening laboratory results for follicle stimulating hormone (FSH) that are within the normal limit for the early follicular phase at the local laboratory
* Is willing and able to comply with the protocol for the duration of the study
* Has voluntarily provided written informed consent and a subject authorization under Health insurance portability and accountability act (HIPAA), prior to any study-related procedure that is not part of normal medical care, with the understanding that the subject could withdraw consent at any time without prejudice to her future medical care

Exclusion Criteria:

* Clinically significant systemic disease
* Known to be infected with Human Immunodeficiency Virus (HIV)
* Known to be infected with Hepatitis C virus
* Known to test positive for Hepatitis B surface antigens
* Any medical condition, which, in the judgment of the Investigator and Sponsor, may interfere with the absorption, distribution, metabolism or excretion of the study drugs
* Known endometriosis Grade III-IV (American society of reproductive medicine [ASRM] classification)
* Uni- or bilateral hydrosalpinx
* Any contraindication to being pregnant and/or carrying pregnancy to term
* Any previous ART cycle indicating a poor response to gonadotropin stimulation (defined as retrieval of three oocytes or less)
* If, in a previous ART attempt, there are no motile sperm before or after the sperm processing with ejaculated, epididymal, testicular, fresh or frozen/thawed spermatozoa
* Three or more previous consecutive ART cycles without a clinical pregnancy
* An extrauterine pregnancy within the last three months before OCP treatment commences
* Abnormal, undiagnosed, gynecological bleeding
* Known allergy or hypersensitivity to human gonadotropin preparations or any other study-related medications
* Known current substance abuse
* Previous participation in this study or simultaneous participation in another clinical trial
* Current smoker

Ages: 18 Years to 39 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 185 (Actual)
Dates: Start 2003-09; Primary Completion 2004-05 (Actual); Study Completion 2004-05 (Actual)

PRIMARY OUTCOMES:
Percentage of subjects without premature luteinizing hormone (LH) surge | r-hCG administration day (end of stimulation cycle {approximately 4 days})

SECONDARY OUTCOMES:
Duration of study treatment | Stimulation Day 1 (S1) up to r-hCG administration day (end of stimulation cycle {approximately 4 days})
Total dose of recombinant human follicle stimulating hormone/human menopausal gonadotropin (r-hFSH/hMG) administered | Stimulation Day 1 (S1) up to r-hCG administration day (end of stimulation cycle {approximately 4 days})
Duration of gonadotropin therapy | Stimulation Day 1 (S1) up to r-hCG administration day (end of stimulation cycle {approximately 4 days})
Number of follicles greater than or equal to (>=) 14 millimeter (mm) on day of recombinant human chorionic gonadotropin (r-hCG) administration | r-hCG administration day (end of stimulation cycle {approximately 4 days})
Number of oocytes retrieved | Ovum pick-up (OPU) day (34-38 hours post r-hCG administration day [end of stimulation cycle {approximately 4 days}])
Number of mature oocytes retrieved | OPU day (34-38 hours post r-hCG administration day [end of stimulation cycle {approximately 4 days}])
Number of fertilized oocytes | Day 1 post OPU day (34-38 hours post r-hCG administration day [end of stimulation cycle {approximately 4 days}])
Number and Quality of Embryos | Day 2-3 post OPU (34-38 hours post r-hCG administration day [end of stimulation cycle {approximately 4 days}])
Implantation rate | Day 35-42 post r-hCG administration day (end of stimulation cycle {approximately 4 days})
Total number of transferred and cryopreserved embryos | Day 2-3 post OPU (34-38 hours post r-hCG administration day [end of stimulation cycle {approximately 4 days}])
Percentage of subjects with clinical and biochemical pregnancies | Day 35-42 post r-hCG administration day (end of stimulation cycle {approximately 4 days})
Quality of Life assessed by Short Form- 36 (SF-36) Questionnaire | Stimulation Day 1 (S1) and Day 15-18 post r-hCG administration (end of stimulation cycle {approximately 4 days})

CONTACTS AND LOCATIONS:
Overall Officials: Eduardo Kelly, MD, MBA, Study Director — EMD Serono

REFERENCES:
- [Background] Wilcox J, Potter D, Moore M, Ferrande L, Kelly E; CAP IV Investigator Group. Prospective, randomized trial comparing cetrorelix acetate and ganirelix acetate in a programmed, flexible protocol for premature luteinizing hormone surge prevention in assisted reproductive technologies. Fertil Steril. 2005 Jul;84(1):108-17. doi: 10.1016/j.fertnstert.2005.03.016. PMID 16009165
- See also: Study published in Fertility & Sterility 84(1):108-17;2005 — http://dx.doi.org/10.1016/j.fertnstert.2005.03.016
- See also: Full FDA approved prescribing information can be found here — http://www.fertilitylifelines.com